CLINICAL TRIAL: NCT02139293
Title: Functional Mapping of Auricular Vagal Stimulation Points on Cardiovascular Parameters in Healthy Subjects - Pilot Study
Brief Title: Pilot Study - Auricular Vagus Nerve Stimulation Effects on Cardiovascular Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Vienna University of Technology (Other)
Responsible Party: Principal Investigator, Dr. Jozsef Constantin Széles, Dr.med., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PS 02/2014
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Modulation of Cardiovascular Parameters and Sympathovagal Balance in Healthy Subjects
Keywords: vagus nerve stimulation effects on heart rate variability and peripheral blood perfusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- auricular vagus nerve stimulation (Experimental): Study participants (healthy) are treated with auricular vagus nerve stimulation using five needle electrodes connected to an electrical stimulation device (PrimeStim). After acclimatization the stimulation is turned on for 20 minutes followed by 20 minutes of paused stimulation, 20 minutes of stimulation, and 10 minutes paused stimulation. This intervention is repeated on four consecutive days, whereas at each intervention only one of the four stimulation points (and one fixed reference point) is stimulated. Needle electrodes are applied at each study visit.
  Stimulation points in the auricle are stimulated in random order. One stimulation pattern is tested. Stimulation amplitudes are adjusted with respect to a distinct but comfortable sensation at the auricle.
  During the described protocol various biosignals are continuously recorded, including ECG, respiration, blood perfusion, oxygen saturation, transcutaneous oxygen tension, blood pressure and skin temperature.
  Interventions: Device: PrimeStim

INTERVENTIONS:
Device: PrimeStim — Intermittent auricular vagus nerve stimulation at different ear points

SUMMARY:
The purpose of this pilot study is to evaluate the effect of auricular autonomous nervous system stimulation on cardiovascular parameters and sympathovagal balance in healthy subjects. It is investigated if auricular vagal nerve stimulation affects heart rate variability as well as peripheral local blood perfusion, and if this effect depends on the site of stimulation in the auricle, whereas four distinct stimulation points are tested.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 20 to 50 years

Exclusion Criteria:

* participation in a clinical trial in the last 5 weeks
* diseases which may affect the autonomous nervous system (e.g., diabetes mellitus)
* confounding medical treatment with known effects on the autonomous nervous system (e.g., beta blocker)
* drug abuse
* active implanted devices
* pregnancy or nursing

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change in heart rate variability (HRV) related to stimulation site in the auricle | within 4 days of intervention, at each day of intervention from baseline to stimulation and pause cycles
  Heart rate variability will be assessed as, e.g., standard deviation in heart rate over a time window of 5 minutes (2.5 minutes overlap), total power or low to high frequency power.
  Changes in assessed heart rate variability parameters will be assessed and compared between subjects with respect to stimulation site using statistical tests.
change in local blood perfusion index (BPI) related to stimulation site in the auricle | within 4 days of intervention, at each day of intervention from baseline to stimulation and pause cycles
  Blood perfusion index at the foot will be assessed as peak-peak amplitude (systolic to diastolic) divided by the mean signal value of optically measured blood perfusion.
  Changes in mean value and standard deviation of local blood perfusion index will be assessed and compared between subjects with respect to stimulation site using statistical tests.

SECONDARY OUTCOMES:
Change of local BPI in upper and lower extremities | within 4 days of intervention, at each day of intervention from baseline to stimulation and pause cycles
  Local BPI is assessed using optical sensors on the foot and the finger of participants.
  Changes in mean value of BPI are analyzed using statistical tests.
Changes in blood pressure | within 4 days of intervention, at each day of intervention from baseline to stimulation and pause cycles
  Blood pressure is continuously measured using inflatable finger cuffs.
Changes in respiratory activity | within 4 days of intervention, at each day of intervention from baseline to stimulation and pause cycles
  Respiratory activity is monitored using a respiratory belt.
Changes in oxygen saturation of the toe | within 4 days of intervention, at each day of intervention from baseline to stimulation and pause cycles
Changes in partial transcutaneous oxygen pressure of the forefoot | within 4 days of intervention, at each day of intervention from baseline to stimulation and pause cycles
Changes in foot skin temperature | within 4 days of intervention, at each day of intervention from baseline to stimulation and pause cycles
Changes of C reactive protein- and leukocyte-concentration in serum | at screening and at the last day of intervention
Tolerance of stimulation | at each day of intervention at the stimulation cycles
  Tolerance of stimulation is assessed by free survey.
Perception of Stimulation | at each day of intervention at the stiumulation cycles
  Perception of stimulation is assessed by free survey.
Adverse effects of stimulation | within 4 days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jozsef C Széles, Dr.med., Principal Investigator — University Clinic for Surgery, Department of Transplantation, Medical University Vienna
Locations (1):
- University Clinic for Surgery, Department of Transplantation, Medical University Vienna, Vienna, Austria